CLINICAL TRIAL: NCT06254911
Title: Window of Opportunity Study of Pre-Operative Atezolizumab (ANTI PD-L1 ANTIBODY) for Patients With Resectable HPV Related Oropharyngeal Squamous Cell Carcinoma (OPSCC)
Brief Title: Pre-operative Atezolizumab in Patients With Resectable, Human Papillomavirus Related Oropharyngeal Carcinoma
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Institutional Review
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Nabil F. Saba, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004678; NCI-2023-01367 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00004678 (Other: Emory University Hospital/Winship Cancer Institute); WINSHIP5730-22 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2024-01-09; First posted 2024-02-12 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Oropharynx Cancer, Stage I
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — atezolizumab; Neck Dissection; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Atezolizumab) (Experimental): Patients receive atezolizumab IV while on study. Patients undergo CT scan and MRI throughout the study. Patients may undergo tumor biopsy while on study.
  Interventions: Biological: Atezolizumab; Procedure: Transoral Surgery with cervical lymphadenctomy (neck dissection); Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Biological: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
Procedure: Transoral Surgery with cervical lymphadenctomy (neck dissection) — Undergo definitive surgical treatment to remove cancer from the tonsil or tongue base combined with removal of the at risk lymph nodes in the neck
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging

SUMMARY:
This phase II trial tests how well atezolizumab works in treating patients with human papillomavirus (HPV) related oropharyngeal squamous cell carcinoma that is able to be removed with surgery (resectable). Immunotherapy with atezolizumab, may include changes in the body's immune system and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety tolerability of 2 doses of single agent atezolizumab in HPV-driven oropharyngeal squamous cell carcinoma (OPSCC).

II. To determine the pathologic response to 2 doses of single agent atezolizumab in HPV-driven OPSCC.

SECONDARY OBJECTIVES:

I. To evaluate the event free survival at 2 years after treated with this approach followed by pathologic directed adjuvant therapy.

EXPLORATORY EFFICACY OBJECTIVES:

I. The exploratory efficacy objective for this study is to evaluate the efficacy of atezolizumab compared with control (previously studied and published in Nature) on the basis of the following endpoints:

Ia. Determine a biomarker profile of responders versus non-responders to atezolizumab by examining the following biomarkers in the tissue and blood.

Ib. Confirm that PD-1 blockade with atezolizumab will result in an effective proliferation and differentiation PD1+, TCF1+ stem like tumor infiltrating lymphocytes (TILs) in the tumor microenvironment (TME) of patients in HPV-driven OPSCC (correlate these findings with pathologic response).

Ic. Study the temporal differentiation and migration of effector-like cells and their correlation with evidence of pathologic response and tumor immune infiltration.

Id. Correlate these findings with evidence of response using circulating tumor deoxyribonucleic acid (ctDNA) in the peripheral blood.

Ie. Examine the B-cell antigen specific cell (ASC) infiltration and characteristics in the TME of patients and correlate these findings with clinical and pathologic responses.

OUTLINE:

Patients receive atezolizumab intravenously (IV) while on study. Patients undergo computed tomography (CT) scan and magnetic resonance imaging (MRI) throughout the study. Patients may undergo tumor biopsy while on study.

ELIGIBILITY:
Inclusion Criteria:

* The subject is >= 18 years old on the day of consent
* Sexually active subjects (men and women) must agree to use medically accepted barrier methods of contraception (eg, male or female condom) during the course of the study and for 5 months after the last dose of study drug(s), even if oral contraceptives are also used. All subjects of reproductive potential must agree to use both a barrier method and a second method of birth control during the course of the study and for 5 months after the last dose of study drug(s).
* Female subjects of childbearing potential must not be pregnant at screening. Females of childbearing potential are defined as premenopausal females capable of becoming pregnant (ie, females who have had any evidence of menses in the past 12 months, with the exception of those who had prior hysterectomy). However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, low body weight, ovarian suppression or other reasons.
* A male participant must agree to use a contraception as detailed in this protocol during the treatment period and for at least during the active treatment plus an additional 90 days (a spermatogenesis cycle) for study treatments with evidence of genotoxicity at any dose] after the last dose of study treatment and refrain from donating sperm during this period.
* The subject has a histologic or cytologic diagnosis of squamous cell carcinoma of the oropharynx, Stage 1 (T1/2 N1) Squamous Cell Carcinoma of the oropharynx associated with HPV as determined by p16 protein expression using immunohistochemistry (IHC) performed by a clinical laboratory improvement act (CLIA) approved laboratory.
* Patients must not have evidence of extensive or "matted/ fixed" pathologic adenopathy on preoperative imaging.
* The subject has had an assessment of all known disease sites eg, by computerized tomography (CT) scan, magnetic resonance imaging (MRI), bone scan or positron emission tomography (PET)/CT scan as appropriate, within 28 days before the first dose of therapy
* The subject is capable of understanding and complying with the protocol requirements and has signed the informed consent document
* Criteria related to comparator drug or background therapy, if applicable: No prior radiation above the clavicles. Patients with a history of a curatively treated malignancy must be disease-free for at least two years prior to entry on study except for carcinoma in situ of cervix, melanoma in-situ (if fully resected), and/or non-melanomatous skin cancer
* Age >= 18 years at time of signing Informed Consent Form
* Ability to comply with the study protocol
* Histologically or cytologically confirmed p16+ HPV-driven OPSCC
* Availability of a representative tumor specimen for exploratory biomarker research
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (1500/GL) without granulocyte colony-stimulating factor support obtained within 14 days prior to initiation of study treatment
* Lymphocyte count >= 0.5 x 10^9/L (500/GL) obtained within 14 days prior to initiation of study treatment
* Platelet count >= 100 x 10^9/L (100,000/GL) without transfusion obtained within 14 days prior to initiation of study treatment
* Hemoglobin >= 90 g/L (9 g/dL) obtained within 14 days prior to initiation of study treatment.

  * Patients may be transfused to meet this criterion
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase (ALP) =< 2.5 x upper limit of normal (ULN), obtained within 14 days prior to initiation of study treatment with the following exceptions:

  * Patients with documented liver metastases: AST and ALT =< 5 x ULN
  * Patients with documented liver or bone metastases: ALP =< 5 x ULN
* Serum bilirubin =< 1.5 x ULN obtained within 14 days prior to initiation of study treatment with the following exception:

  * Patients with known Gilbert disease: serum bilirubin =< 3 x ULN
* Serum creatinine =< 1.5 x ULN obtained within 14 days prior to initiation of study treatment
* Serum albumin >= 25 g/L (2.5 g/dL) obtained within 14 days prior to initiation of study treatment
* For patients not receiving therapeutic anticoagulation: international normalization ratio (INR) or activated partial thromboplastin time (aPTT) =< 1.5 x ULN obtained within 14 days prior to initiation of study treatment
* For patients receiving therapeutic anticoagulation: stable anticoagulant regimen
* Negative human immunodeficiency virus (HIV) test at screening, with the following exception: patients with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4 count >= 200/uL, and have an undetectable viral load
* Negative hepatitis B surface antigen (HBsAg) test at screening
* Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV ribonucleic acid (RNA) test at screening. The HCV RNA test must be performed for patients who have a positive HCV antibody test

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from study entry:

* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

  * Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
  * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
* Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

  * Rash must cover < 10% of body surface area
  * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
  * There has been no occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Active tuberculosis
* History of leptomeningeal disease
* Uncontrolled tumor-related pain
* Patients requiring pain medication must be on a stable regimen at study entry
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently) Patients with indwelling catheters (e.g., PleurX) are allowed.
* Uncontrolled or symptomatic hypercalcemia (ionized calcium >1.5 mmol/L, calcium >12mg/dL or corrected serum calcium >ULN)
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia, or any active infection that could impact patient safety.
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* History of malignancy must have been treated with curative intent and must be disease free for 1 year prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as adequately treated carcinoma in situ of the cervix or non-melanoma skin carcinoma
* Prior allogeneic stem cell or solid organ transplantation
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab
* Current treatment with anti-viral therapy for HBV
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

  * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study.
  * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 5 months after the final dose of study treatment. Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment
* Glomerular filtration rate < 29 mL/min/1.73 m^2 as calculated through use of the Chronic Kidney Disease Epidemiology Collaboration equation
* An ANC < 1.5 x 10^9/L (1500/GL) with one exception:

  * Patients with benign ethnic neutropenia (BEN): ANC < 1.3 x 10^9/L (1300GL) BEN (also known as constitutional neutropenia) is an inherited cause of mild or moderate neutropenia that is not associated with any increased risk for infections or other clinical manifestations. BEN is referred to as ethnic neutropenia because of its increased prevalence in people of African descent and other specific ethnic groups

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2026-12-16 (Estimated); Study Completion 2026-12-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | From the first dose of study drug to 30 days after the last dose of the study drug
Pathologic response | After cycle 2 (each cycle is 21 days) and prior to surgery (for ctDNA changes) and on final pathologic analysis 14 days after surgery
  Defined as human papillomavirus (HPV) circulating tumor deoxyribonucleic acid (ctDNA) level by interval change in pre- versus post-treatment HPV ctDNA level.
Event-free survival (EFS) | From the first administration of atezolizumab to date of recurrence, death or up to 2 years
  Defined as the time from the first administration of 2 doses of single agent atezolizumab to the date of recurrence or death due to any cause, and patients who did not experience recurrence or death will be censored at the last evaluable disease assessment. The EFS distribution will be estimated by constructing a Kaplan-Meier curve with estimation of 2-year EFS rate and 95% CI.

SECONDARY OUTCOMES:
Association of biomarkers with pathological response status | Up to 2 years
  Tested by two-sample t-test with p-value being adjusted for multiple testing using Tukey's method. The longitudinal change pattern (e.g., increase or decrease) of a biomarker over the course of treatment will be captured and described graphically. Both change pattern and baseline values of a biomarker will be used to associate with EFS using Cox proportional hazard model to see whether it can be predictive or prognostic. The predictive performance will be summarized as Uno's C-index and 95% CI for discrimination. Multivariable model in logistic regression or Cox regression will be further considered to control possible confounding effects in the correlation due to the nature of observational trial and correlative design.

CONTACTS AND LOCATIONS:
Overall Officials: Nabil F. Saba, MD, FACP, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University Hospital Midtown, Atlanta, Georgia, United States